CLINICAL TRIAL: NCT07102823
Title: Clinical Registry for the Characterization of the 'Pulmonary Vascular Phenotype' in Patients With Chronic Obstructive Pulmonary Disease - a Retrospective Multi-center Data Analysis
Brief Title: Clinical Registry for the Characterization of the 'Pulmonary Vascular Phenotype' in Patients With Chronic Obstructive Pulmonary Disease
Acronym: COPD-PH
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 35-272ex22/23
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Pulmonary Hypertension
Keywords: pulmonary hypertension; chronic obstructive pulmonary disease; right heart catheterization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Registry of COPD (Chronic Obstructive Pulmonary Disease) patients who underwent right heart catheterization (RHC) and full clinical evaluation for pulmonary hypertension

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD
* right heart catheterization including mPAP (Mean Pulmonary Artery Pressure), PVR (Pulmonary Vascular Resistance), PAWP (Pulmonary Artery Wedge Pressure), CO (cardiac output)
* age >= 18 years

Exclusion Criteria:

* pediatric patients
* no COPD or no RHC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients who underwent RHC
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Severe Pulmonary Hypertension (PH) | at inclusion
  pulmonary vascular resistance > 5 WU (Wood Units)
all-cause mortality | Until 2026
  all-cause mortality

CONTACTS AND LOCATIONS:
Locations (3):
- Medical University of Graz, Graz, Austria
- University of Zurich, Zurich, Switzerland
- University of Sheffield, Sheffield, United Kingdom